CLINICAL TRIAL: NCT02872480
Title: The Effect of ACTIVE Training in Improving Clinical Outcomes in Healthy and Acutely Concussed College-aged Participants
Brief Title: Acute Concussion Therapy Intervention Training in Healthy and Concussed Participants
Acronym: ACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-2387; 16-2829 (Other Grant/Funding Number: American College of Sports Medicine)
Record Dates: First submitted 2016-07-27; First posted 2016-08-19 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Cerebral Concussion
Keywords: Concussion; Exercise
MeSH Terms: conditions — Brain Concussion; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACTIVE Training (Experimental): Healthy participants will be progressed from 60-80% of their VO2max as determined by the progressive exercise test over the course of 6 30-minute training sessions. Concussed participants will begin 30-minute training sessions at 60% of the VO2 achieved at symptom exacerbation of the exercise test. Intensity will be progressed as tolerated by the participant and training sessions will continue until the participant is asymptomatic for 24 consecutive hours (total number of sessions variable based on clinical recovery).
  Interventions: Other: ACTIVE Training
- Control (No Intervention): Healthy controls will be asked to follow their normal routine for rest and physical activity. Concussed controls will be asked to follow the guidance for rest and activity as prescribed by the physicians and athletic trainers overseeing their clinical care.

INTERVENTIONS:
Other: ACTIVE Training — Participants will be asked to complete aerobic exercise on a stationary bike during 30-minute sessions. Intensity will progress under a standard procedure for healthy participants (60-80% of VO2max) and as tolerated by concussed participants (starting at 60% of symptom exacerbation).
  Arms: ACTIVE Training

SUMMARY:
Healthy (non-injured) and concussed college-aged participants will complete two testing sessions that include (1) clinical symptom, balance, and cognitive evaluations and (2) a progressive exercise session to establish symptom exacerbation or maximal exercise capacity. Individuals randomized to the control group will receive no intervention between sessions, while individuals randomized to the intervention group will complete 30 minutes of stationary bike exercise at least 3 days/week.

DETAILED DESCRIPTION:
Healthy and concussed participants will be randomized to ACTIVE training (intervention) or control (no intervention) groups. Participants, regardless of group assignment, will receive clinical symptom, balance, and cognitive evaluations as well as a progressive exercise assessment at study outset. Concussed participants will enroll into the study within three days of injury and study participation will termination following 24 consecutive hours with no reported concussive symptoms. Healthy participants will have arbitrary start dates and will terminate the study 10-14 days later to approximate the general length of concussion recovery and, therefore, make the time between session in the healthy and concussed cohorts as equivalent as possible. Participants in the intervention group will complete stationary cycle ergometer workouts for 30 mins at least 3 days per week between testing sessions. Healthy participants will complete six ACTIVE training sessions, while concussed participants will complete ACTIVE training at least three days per week until asymptomatic. Concussed control participants will follow physician guidelines for rest and activity, while healthy control participants will be asked to follow their typical routines for rest and activity. Participants will repeat the identical testing session assessments prior to study termination.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having a concussion by a physician within three days of study enrollment (concussed participants only)
* Glasgow Coma Scale >13 (concussed participants only)
* Participants must be active, which is defined as 30 or more minutes of moderate to vigorous physical activity 3 or more days per week. All healthy participants must met this definition and concussed participants should have met this definition prior to injury.
* Good cardiovascular health (subject to approval from study physician)

Exclusion Criteria:

* Recreational drug use over the course of study participation
* Associated injuries (broken bones, etc.) that would limit the ability to successfully complete ACTIVE training
* For healthy participants, no history of concussion within the last year
* For concussed participants, skull fracture or brain bleed at time of the injury
* UNC Varsity athletes

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Average Days to Recovery | Assessed every 24 hours from baseline to study termination for each participant (approximately 10-14 days)
  Average number of days from injury to recovery (recovery is defined as full clearance by physician)

SECONDARY OUTCOMES:
Average Change in Mental Status | Each participant will complete the SAC at baseline (first testing session) and recovery (full clearance by physician)- approximately 10-14 days apart
  SAC Total Score (Out of 30 possible points; combination of scores from orientation (5), immediate memory (15), concentration (5), and delayed memory (5) sections; higher scores are indicative of better results)
Average Changed in Balance | Each participant will complete the BESS at at baseline (first testing session) and recovery (full clearance by physician)- approximately 10-14 days apart
  BESS Total Score (Participants are given errors for positions of poor postural control; out of 60 points; higher scores are indicative of poorer performance)
Average Change in Cognition | Each participant will complete CNS at at baseline (first testing session) and recovery (full clearance by physician)- approximately 10-14 days apart
  CNS Composite Score (percentile of participant's overall achievement on a computerized neurocognitive test; higher percentiles indicate better performance)
Average Change in Near-Point Convergence | Each participant will complete the VOMS at at baseline (first testing session) and recovery (full clearance by physician)- approximately 10-14 days apart
  Near-point convergence distance (average distance- over three trials- of convergence during vision, higher scores indicate poorer convergence)
Average Change in Concussive Symptoms | Healthy participants will complete the GSC at at baseline (first testing session) and recovery (full clearance by physician)- approximately 10-14 days apart
  GSC Total Score (incorporates presence and severity for a total score on 27-items, each item rated from 0 (not present) to 6 (severe); higher scores indicate worse symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth F Teel, M.S., Principal Investigator — University of North Carolina, Chapel Hill; Jason P Mihalik, Ph.D., Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teel EF, Register-Mihalik JK, Appelbaum LG, Battaglini CL, Carneiro KA, Guskiewicz KM, Marshall SW, Mihalik JP. Randomized Controlled Trial Evaluating Aerobic Training and Common Sport-Related Concussion Outcomes in Healthy Participants. J Athl Train. 2018 Dec;53(12):1156-1165. doi: 10.4085/1062-6050-7-18. Epub 2018 Dec 18. PMID 30562056